CLINICAL TRIAL: NCT00765154
Title: Phase IV, Two-arm, Open-label, Single-centre Randomised Pilot Study to Assess the Feasibility of Immediate or Deferred Switching of HIV-infected Individuals Intolerant of Efavirenz, Ritonavir-boosted Lopinavir or Ritonavir-boosted Darunavir
Brief Title: NNRTI/PI Toxicity Switch to Darunavir Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties in recruitment due to a change in the nature of practice.
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Mark Nelson, St Stephens Aids Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 028
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: HIV
MeSH Terms: interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Immediate switch from NNRTI/PI to DRV/r
  Interventions: Drug: darunavir
- Group 2 (Active Comparator): Switch after 10 weeks from NNRTI/PI to DRV/r
  Interventions: Drug: ritonavir

INTERVENTIONS:
Drug: darunavir — two 400mg tablets (800mg) once daily
  Other Names: TMC114; Trade Name: Prezista
  Arms: Group 1
Drug: ritonavir — one 100mg capsule once daily
  Other Names: Trade Name: Norvir
  Arms: Group 2

SUMMARY:
The purpose of the study is to examine the effects of switching from antiretroviral combinations that includes efavirenz (Sustiva®), lopinavir/ritonavir (Kaletra®) or atazanavir/ritonavir (Reyataz®/Norvir®) in individuals experiencing side effects from one of these agents, and replacing these with a new HIV medication called Darunavir also given with ritonavir (Norvir®).

The study will primarily investigate the effect of change in medication on the subjects viral load (the levels of the HIV virus in the blood), on immunological parameters (CD4 count) and on other safety parameters (such as cholesterol) and also quality of life.

DETAILED DESCRIPTION:
The advent of highly active antiretroviral therapy (HAART) has revolutionised the treatment of HIV disease, with both patients and physicians enjoying the marked reductions in HIV related morbidity and mortality. However, as long term therapeutic success has become a realistic goal of treatment, there are increasing reports of toxicities associated with therapy.

Indeed since the advent of HAART the major reason for change in therapy has not been a lack of efficacy associated with drug regimens but the toxicity associated with individual agents. Although the potential adverse events associated with antiretrovirals are manifold there are signature treatment-limiting toxicities associated with particular agents such as EFV and CNS/neuropsychiatric adverse events, LPV/r and gastrointestinal toxicity and ATV/r and jaundice.

A recent study performed at the Chelsea and Westminster hospital showed that 61% of regimen switches were due to toxicity and the majority of these occurred after 12 weeks of therapy.

Darunavir is a recently licensed protease inhibitor which requires ritonavir boosting.Currently DRV/r is licensed for use in treatment-experienced individuals. In triple-class experienced patients ritonavir boosted darunavir has been associated with greater viral load reductions when combined with optimized background (OB) than OB alone. A study of PI experienced patients randomized to receive Kaletra or ritonavir boosted darunavir with optimised background therapy showed significantly higher rates of virological suppression in the DRV/r arm; rates of toxicities were similar overall but less diarrhoea in the DRV/r than the Kaletra arm. Darunavir is licensed twice daily and has a high barrier to the development of resistance. DRV/r dosed at 800/100mg once daily has been compared with LPV/r in treatment-naïve subjects. DRV/r was non-inferior to LPV/r overall and performed significantly better than LPV once daily and in subjects with a high baseline viral load. DRV/r and LPV/r have also been compared head to head in 'early'treatment-experienced patients (failing first or second line therapy but LPV-naive). Overall DRV/r exhibited superiority to LPV/r with 77% and 67% achieving viral suppression to less than 50 copies/ml by intent-to-treat analysis respectively (95% confidence interval for the difference 2-17%; p <0.0001). Animal studies have shown a low risk of teratogenesis associated with DRV.

This study aims to investigate whether substitution of NNRTI/PI with ritonavir boosted darunavir leads to resolution of toxicity associated with these drugs, continued virological suppression and immunological reconstitution and whether this is associated with an improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected as documented by a licensed HIV-1 antibody ELISA test
* Subject is currently on an antiretroviral regimen comprising of at least three licensed antiretroviral agents including efavirenz, ritonavir-boosted lopinavir or ritonavir-boosted atazanavir
* Subject is virologically suppressed with a viral load < 50 copies/ml
* Subject has a CD4+ count above 50 cells/ml
* If subject is a female of childbearing potential, she must agree to use a double barrier method of contraception
* No previous exposure to darunavir

Exclusion Criteria:

* Pregnant or lactating women
* Any female of childbearing potential not using effective birth control methods or not willing to continue practicing these birth control methods during the trial and for at least 30 days after the end of the trial (or after last intake of investigational ARVs)
* Heterosexually active male subject not using effective birth control methods or not willing to continue practicing these birth control methods during the trial and until 30 days after the end of the trial (or after last intake of investigational ARVs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The improvement of NNRTI/PI associated toxicity after 4 weeks of therapy with ritonavir boosted darunavir. | 20 days

SECONDARY OUTCOMES:
Viral load suppression below 50 copies/ml post switch | between 20 and 60 days
Viral load < 400 copies/ml post switch | between 20 and 60 days
Toxicity | 60 days
Health related quality of life questionnaires | Baseline, 20 and 60 days
Changes in fasting triglycerides post switch | 20 days and 60 days
Adherence as measured via questionnaire | baseline, 20 days and 60 days
Tolerability as measured by tolerability index questionnaire (HIV patients symptoms profile | baseline, 20 days and 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom